CLINICAL TRIAL: NCT01075932
Title: The Cognitive And Cerebral Hemodynamic Effects Of DHA-Rich Fish Oil: A Dose-Ranging Study
Brief Title: Effects of Docosahexaenoic Acid (DHA)-Rich Fish Oil on Cerebral Haemodynamics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Ginsana SA (Other)
Responsible Party: Philippa Jackson, Northumbria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 16N2
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2010-02-25 (Estimated); Status verified 2010-02

CONDITIONS: Cerebral Blood Flow; Cognitive Function
Keywords: cerebral blood flow; NIRS; n-3 PUFAs; fish oil; cognitive function

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 g DHA-rich fish oil (Active Comparator): 1 g DHA-rich fish oil containing 450 mg DHA + 90 mg EPA plus 1 g olive oil
  Interventions: Dietary Supplement: DHA-rich fish oil
- 2 g DHA-rich fish oil (Active Comparator): 2 g DHA-rich fish oil containing 900 mg DHA + 180 mg EPA
  Interventions: Dietary Supplement: DHA-rich fish oil
- Placebo (Placebo Comparator): 2 g olive oil
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: DHA-rich fish oil — Either 1 g or 2 g DHA-rich fish oil taken daily for 12 weeks. Participants in the 1 g group will also consume 1 g olive oil placebo capsules per day to maintain double blind.
  Arms: 1 g DHA-rich fish oil; 2 g DHA-rich fish oil
Dietary Supplement: Placebo — 2 g placebo (olive oil) taken daily for 12 weeks
  Arms: Placebo

SUMMARY:
DHA has previously been shown to increase regional cerebral blood flow response to tactile stimulation in aged monkeys; modulation of cerebral blood flow in humans has yet to be demonstrated. Given that the brain relies on a constant supply of blood-borne metabolic substrates (e.g. glucose, oxygen), increasing regional cerebral blood flow may also have an impact on cognitive function. The current study aims to investigate the effects of two doses of DHA-rich fish oil on task-related cerebral hemodynamic response and cognitive performance in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female
* 18-35 years
* Healthy
* No herbal supplements/prescription medications (excl. contraceptive pill)
* Non smoker
* Native English speaker

Exclusion Criteria:

* consumes oily fish
* takes omega-3 supplement
* food allergies to treatment ingredients

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2009-04; Primary Completion 2009-05 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Cerebral blood flow | 12 weeks
  Cerebral blood flow will be assessed using Near Infrared Spectroscopy while participants complete a series of cognitive tasks.

SECONDARY OUTCOMES:
Cognitive function | 12 weeks
  Cognitive function will be assessed using a series of tasks that evaluate working memory, attention and executive function.

CONTACTS AND LOCATIONS:
Overall Officials: Philippa A Jackson, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

REFERENCES:
- [Derived] Jackson PA, Reay JL, Scholey AB, Kennedy DO. Docosahexaenoic acid-rich fish oil modulates the cerebral hemodynamic response to cognitive tasks in healthy young adults. Biol Psychol. 2012 Jan;89(1):183-90. doi: 10.1016/j.biopsycho.2011.10.006. Epub 2011 Oct 19. PMID 22020134
- See also: Brain, Performance and Nutrition Research Centre, Northumbria University — http://www.nutrition-neuroscience.co.uk/